CLINICAL TRIAL: NCT06694519
Title: Effectiveness of Radiofrequency and Exercise-based Rehabilitation on Symptoms Associated With Pelvic Floor Dysfunction in Breast Cancer Patients.
Brief Title: Radiofrequency and Exercise-based Rehabilitation on Symptoms Associated With Pelvic Floor Dysfunctions in Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SERGIO MONTERO NAVARRO (Other)
Collaborators: Cardenal Herrera University (Other); CAPENERGY MEDICAL, SL (Industry)
Responsible Party: Sponsor-Investigator, SERGIO MONTERO NAVARRO, Clinical Professor, Cardenal Herrera University
Organization: Cardenal Herrera University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: CEEI24/540
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Genitourinary Syndrome; Radiofrequency; Physical Exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Pain Measurement

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temperature after apply RF in capacitive electrical transfer mode (Capernergy® device model C500) (Experimental): It is a device designed mainly to address dysfunctions in the urogynecological area, where the increase in tissue temperature is regulated by a temperature sensor, with 3 frequencies (0.8MHz, 1MHz and 1.2 MHz) that will allow different tissue depths to be addressed, and a power of 310w. This device consists of two electrodes: an active capacitive electrode to be placed in the vaginal area with a probe cover and water-soluble gel and another dispersive electrode or return plate to be positioned in the lumbosacral region.
  Interventions: Device: manometry through the PHENIX series device (model: PHENIX LIBERTY; manufacturer: ELECTRONIC CONCEPT LIGNON INNOVATION, Montpelier, France).; Diagnostic Test: PFIQ-20 questionnaire (Pelvic Floor Impact Questionnaire Short Form); Diagnostic Test: ICIQ-SF (International Consultation on Incontinence Questionnaire - Short Form); Diagnostic Test: Sandvik's test; Diagnostic Test: vaginal health index (VHI); Diagnostic Test: Visual analogue scale (VAS); Diagnostic Test: Body Image Scale (S-BIS); Diagnostic Test: Likert's scale questionnaire; Diagnostic Test: Oxford's Scale; Diagnostic Test: Sexual function and self-esteem
- PFMT (Experimental): The PFMT will consist of a targeted programme, with a protocol of CORE and pelvic floor exercises established based on the assessment of the patients' strength, endurance and fatigue, with a frequency of twice a week led by a physiotherapist and a duration of 45 minutes each day and a period of 16 weeks.It will be carried out in groups of 8 people and accompanied by a physiotherapist experienced in therapeutic exercise.
  Each session will consist of exercises to activate the pelvic floor muscles in isolation and in association with the CORE muscles, both static and dynamic.
  Interventions: Device: manometry through the PHENIX series device (model: PHENIX LIBERTY; manufacturer: ELECTRONIC CONCEPT LIGNON INNOVATION, Montpelier, France).; Diagnostic Test: PFIQ-20 questionnaire (Pelvic Floor Impact Questionnaire Short Form); Diagnostic Test: ICIQ-SF (International Consultation on Incontinence Questionnaire - Short Form); Diagnostic Test: Sandvik's test; Diagnostic Test: vaginal health index (VHI); Diagnostic Test: Visual analogue scale (VAS); Diagnostic Test: Body Image Scale (S-BIS); Diagnostic Test: Likert's scale questionnaire; Diagnostic Test: Oxford's Scale; Diagnostic Test: Sexual function and self-esteem

INTERVENTIONS:
Device: manometry through the PHENIX series device (model: PHENIX LIBERTY; manufacturer: ELECTRONIC CONCEPT LIGNON INNOVATION, Montpelier, France). — For this manometry the air probe, connected to the Phenix biofeedback system, covered by a latex probe cover lubricated with gel, will be used. In the procedure, the labia majora are opened with one hand and slowly rotated into the vagina while holding the back of the manometric probe with the other hand. Basal tone in g will be measured prior to pelvic floor muscles force measurements. The manometry probe will extract pelvic floor pressure signals by measuring both your basal tone and the maximum pressure held for 10 seconds in three measurements, the average of the three being calculated at the command, 'contract as hard as you can for as long as possible'.
Diagnostic Test: PFIQ-20 questionnaire (Pelvic Floor Impact Questionnaire Short Form) — This questionnaire allows assessment of the impact of urinary symptoms, colo-rectal-anal symptoms and genital prolapse symptoms. This questionnaire will also be used as an inclusion criterion, to homogenise the characteristics of the population in terms of pelvic dysfunction prior to the intervention, as indicated above.
Diagnostic Test: ICIQ-SF (International Consultation on Incontinence Questionnaire - Short Form) — a four-question self-administered questionnaire that identifies individuals with urinary incontinence by assessing frequency, severity and impact on quality of life. It is composed of five questions assessing frequency, severity and impact of UI, plus a set of eight self-diagnostic items related to UI situations experienced by patients. The maximum sum of the response values indicates a score of 21 points, referring to the high impact of UI on an individual's life.
Diagnostic Test: Sandvik's test — It provides information on the severity of the UI by means of two questions. The interpretation based on the score is classified as: 1-2 mild UI, 3-6 moderate UI, 8-9 severe UI, 12 very severe UI.
Diagnostic Test: vaginal health index (VHI) — this index consists of a graduated scale from 1 to 5 for each item (vaginal elasticity, fluid volume, pH, epithelial integrity and moisture).Vaginal elasticity ranges from 1 (no elasticity) to 5 (excellent elasticity), assessed by distension of the mucosa on palpation and speculum placement. The volume of fluid, assessed during inspection, varies between 1 (no discharge) and 5 (normal discharge) (white flocculent). The integrity of the epithelium varies between 1 (petechiae already detected on inspection) and 5 (non-friable tissue and normal mucosa). Moisture ranges from 1 (no moisture detected on inspection and presence of inflamed mucosa) to 5 (normal moisture). The pH will be quantified using a pH indicator strip between 0 and 14 (MColorpHast™-PH indicator strips) to be placed directly on the right lateral vaginal wall for one minute, giving 1 point for pH 6.1, 2 for pH 5.6-6.0, 3 for pH 5.1-5.5, 4 for pH 4.7-5.0 and 5 for pH ≤ 4.6. The sum of all items represents the vaginal health
Diagnostic Test: Visual analogue scale (VAS) — This scale allows the intensity of pain described by the patient to be measured with maximum reproducibility between observers. It consists of a horizontal line of 10 centimetres, at the ends of which are the extreme expressions of a symptom. At the left end is the absence or lowest intensity and at the right end the highest intensity. The patient is asked to mark on the line the point that indicates the intensity of the pain during sexual intercourse and it is measured with a millimetres ruler. The intensity is expressed in centimetres or millimetres. The rating will be: 1 Mild pain if the patient scores the pain as less than 3; 2 Moderate pain if the rating is between 4 and 7; 3 Severe pain if the rating is equal to or greater than 8.
Diagnostic Test: Body Image Scale (S-BIS) — It consists of 10 items assessing various dimensions of body image in cancer patients, evaluating: affective, behavioural and cognitive. The items are scored on a four-point scale (0: not at all; 1: a little; 2: quite a lot; 3: a lot) with a maximum possible score of 3 points. The higher the score, the higher the body image problem. Its brevity facilitates rapid assessment in both clinical and research settings. It shows a stable factor structure between samples, and good psychometric properties with high reliability (Cronbach's alpha=0.93), suggesting that it is a suitable and useful measure for assessing body image in breast cancer patients.
Diagnostic Test: Likert's scale questionnaire — five-point Likert scale for satisfaction with treatment to be classified as: 1 (very dissatisfied), 2 (dissatisfied), 3 (no change), 4 (satisfied), 5 (very satisfied). Women who miss any of the RF sessions and/or whose attendance at the face-to-face physiotherapy sessions (RF and/or PFMT) does not reach 80% will be considered as not complying with the study protocol and their participation will be terminated, although they will be included in the analysis (by intention to treat).
Diagnostic Test: Oxford's Scale — It allows the contractile capacity of the pelvic floor muscles to be assessed. It scores from 0 to 5, as follows: if there is no contraction it is 0, if the contraction is very weak it is 1, if the contraction is weak it is 2, if the contraction is moderate/with tension/and maintained it is 3, if the contraction is good and maintains tension with resistance it is 4, and if the contraction is strong and maintains tension against a resistant force it is 5.
Diagnostic Test: Sexual function and self-esteem — The Female Sexual Function Index (FSFI) questionnaire consists of 19 items that assess sexual function over the past 4 weeks and performance in six domains: sexual desire, arousal, lubrication, orgasm, satisfaction and pain. A cut-off point ≤ 26.5 is considered sexual dysfunction and an increase in score is considered an improvement.

SUMMARY:
Breast cancer has a high impact, affecting 2.3 million women worldwide in 2022. In Spain, there were 40,203 new cases in 2023. In addition to the economic and social costs, patients suffer genitourinary dysfunctions due to cancer treatments. Genitourinary Menopausal Syndrome (GUS) affects 50% of menopausal women, with a higher prevalence in women with breast cancer.

This study aims to compare the effectiveness of radiofrequency (RF) and pelvic floor muscle exercise (PFMT) in the treatment of pelvic dysfunction associated with GUS in breast cancer patients. A randomised, double-blind clinical trial will be conducted in collaboration with the Association of Women Affected by Breast Cancer of Elche and Region) and the CEU Cardenal Herrera University. Women diagnosed with breast cancer and pelvic dysfunction will participate, divided into three groups: one will receive PFMT, one will receive RF and one will receive PFMT+RF therapy.

Both techniques are expected to improve the quality of life of patients, where RF could offer additional benefits due to its proven effectiveness in the treatment of vaginal dryness and dyspareunia. The expected results will contribute to more effective and less invasive treatment protocols. The project presented has the potential to positively impact the health and well-being of women with breast cancer, reducing the symptoms associated with the disease and its treatment, and improving their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* women of legal age with a clinical history of breast cancer, who agree to participate in the study and who present pelvic dysfunction assessed by the Pelvic Floor Distress Inventory (PFDI20) ≥ 100
* women survivors of stage 1 and 2 breast cancer
* A medical discharge was granted more than one year ago
* A diagnosis of another type of cancer has not been made.

Exclusion Criteria:

* Having performed PMFT or received RF in the last 12 months
* Use of vaginal oestrogens in the last 6 months
* Systemic hormone therapy in the last 6 months
* Laser therapy in the last 6 months
* Absence of pelvic floor contraction according to the Modified Oxford Scale
* Use of pacemaker
* Use of heart pacemaker, decompensated heart or metabolic diseases, cognitive deficits, peripheral or central neurological disorders, previous surgeries in the pelvic region, skin pathologies or wounds in the treatment area or presence of an active urinary tract and/or vaginal infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
PFDI-20 questionnaire (300 points) | Pre-intervention / a year post-intervention
  This questionnaire assesses the impact over the last 3 months of urinary symptoms (Urinary Impact Questionnaire; UIQ-7), colorectal-anal symptoms (Colorectal-Anal Impact questionnaire, CRAIQ-7) and genital prolapse symptoms (Pelvic Organ Prolapse Impact Questionnaire, POPIQ-7). The maximum possible score is 300 points, with a maximum value of 100 points for each subscale. The higher the score, the greater the negative impact on quality of life.

SECONDARY OUTCOMES:
Age (years) | Pre-intervention
  Subject's age (years)
Sex (female or male) | Pre-intervention
  Subject's sex (female or male)
Body mass index (Kg /m2) | Pre-intervention
  It is a measure of body fat based on height and weight that applies to adult men and women
Pelvic floor muscle strength assessment (oxford scale 0-5 points) | pre-intervention / 15 days post-intervention / 6 months post-intervention / 12 months post-intervention
  If there is no contraction it is rated 0, if the contraction is very weak it is rated 1, if the contraction is weak it is 2, if the contraction is moderate/with tension/and maintained it is 3, if the contraction is good and maintains tension with resistance it is 4, and if the contraction is strong and maintains tension against a resistant force it is 5. In addition, this assessment allows the determination of static muscular endurance, fatiguability or dynamic endurance and maximum muscular strength.
neuromuscular stimulation device and PHENIX LIBERTY manometry (mmHg) | pre-intervention / 15 days post-intervention / 6 months post-intervention / 12 months post-intervention
pH (0-14) | pre-intervention / 15 days post-intervention / 6 months post-intervention / 12 months post-intervention
  The pH will be quantified using a pH indicator strip between 0 and 14 to be placed directly on the right lateral vaginal wall for one minute, giving 1 point for pH 6.1, 2 for pH 5.6-6.0, 3 for pH 5.1-5.5, 4 for pH 4.7-5.0 and 5 for pH ≤ 4.6. The sum of all items represents the vaginal health score, where 25 represents the best vaginal health.

CONTACTS AND LOCATIONS:
Overall Officials: ANA LOZANO, MsC, Principal Investigator — CARDENAL HERRERA - CEU; CEU UNIVERSITIES; CRISTINA ORTS-RUIZ, PhD, Study Director — CARDENAL HERRERA - CEU; CEU UNIVERSITIES; JESÚS SÁNCHEZ-MAS, PhD, Study Director — CARDENAL HERRERA - CEU; CEU UNIVERSITIES
Locations (1):
- Cardenal Herrera - Ceu, Elche, Spain / Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The general data of the subject will be collected (name, age, sex, physical variables and clinical history). You must come to participate in our study with comfortable clothes.
  The personal data are confidential, apply to the protection of personal data. The study will be carried out in accordance with the Declaration of Helsinki and in accordance with current Spanish legislation (Royal Decree 223/2004 and the Biomedical Research Act 2007) and any other thing that may be applicable.
  An alpha-numeric code will be assigned to each participant. The study is double-blind. Only this code will be recorded by the evaluators.
  This study was approved by the Research and Ethics Committee of CEU Cardenal Herrera University (CEEI24/540).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 1 years after the publication of results

REFERENCES:
- [Derived] Salar-Andreu C, Montero-Navarro S, Lozano-Rubio A, Del Rio-Medina S, Botella-Rico JM, Torres-Lacomba M, Benitez-Martinez JC, Sanchez-Mas J, Orts-Ruiz C. Effectiveness of radiofrequency and exercise-based rehabilitation on symptoms associated with pelvic floor dysfunction in breast cancer patients: A study protocol. PLoS One. 2025 Aug 29;20(8):e0330156. doi: 10.1371/journal.pone.0330156. eCollection 2025. PMID 40880350

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT06694519/Prot_SAP_ICF_000.pdf